CLINICAL TRIAL: NCT02180568
Title: Validation Study to Evaluate the Safety and Efficacy of Preoperative Computed Tomography-guided Localization Technique Using Lipiodol for Patients With Ground Glass Opacity Pulmonary Lesions: A Prospective Multicenter Study
Brief Title: Lipiodol Localization for Ground-glass-opacity Minimal Surgery
Acronym: LOGIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Collaborators: Gangnam Severance Hospital (Other); Asan Medical Center (Other); Pusan National University Hospital (Other); Korea University Anam Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Dankook University (Other); Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Jin Hur, professor, Severance Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SEV2013-0740; F015894 (Other Grant/Funding Number: Guerbet Korea)
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Lesion With Ground-glass-opacity
Keywords: Ground-glass-opacity (GGO); Lung localization; Lipiodol; Hook wire; Video assisted thoracic surgery (VATS)
MeSH Terms: interventions — Ethiodized Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lipiodol (Experimental): Lipiodol-guided lung localization technique
  Interventions: Procedure: Lipiodol; Drug: Lipiodol
- Hookwire (Active Comparator): Hookwire-guided lung localization technique
  Interventions: Procedure: Hookwire

INTERVENTIONS:
Procedure: Lipiodol — Lipiodol-guided lung localization technique
  Arms: Lipiodol
Procedure: Hookwire — Hookwire-guided lung localization technique
  Arms: Hookwire
Drug: Lipiodol
  Arms: Lipiodol

SUMMARY:
The study object is to demonstrate the usefulness and safety of lipiodol localization technique for individuals undergoing ground-glass opacity (GGO) Video-assisted thoracic surgery (VATS) resection compared to hook wire localization technique. A total of 250 participants will be enrolled in a 1:1 fashion to Lipiodol or Hook-wire groups. If the aims of this study are achieved, the use of lipiodol localization technique will be widespread their application for localization of non-palpable pulmonary lesions that are indicated for VATS resection.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adult patients ≥ 20 years of age
* Pulmonary lesion with a ground glass opacity(GGO)component of more than 50%
* Patient with lesion size less than 3cm
* Persistence or growth of the established lesion within a three month period
* Patient who are not contraindicated to surgery
* Patients who are willing to sign the informed consent form

Exclusion Criteria:

* Patients with solid pulmonary lesion
* Patients with multiple GGOs need multiple localization
* Patients who are contraindicated to surgery
* Patients who behave in an uncooperative manner
* Unwilling or unable to give informed consent
* Pregnant women

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Procedure success rate | one day
  Procedure success was defined as marking (lipiodol or hook-wire) the GGO lesion within 1 cm without pleural leakage of lipiodol or dislodgement of the hook-wire.

SECONDARY OUTCOMES:
Complication rate | one day
  Procedure-related complications such as pneumothorax, lung hemorrhage, hemoptysis, air-embolism and death
Procedure time | 1 hour
  Total procedure time for lung localization
Surgery time | 12 hours
  Surgery time for obtaining wedge resection specimen
Safety resection margin | 1 hour
  The safety specimen resection margin was categorized either as positive (grossly positive (R2), microscopically positive if tumor was at the inked surface (R1)), or negative (microscopically negative if there was no tumor at the inked surface (R0))

CONTACTS AND LOCATIONS:
Overall Officials: Jin Hur, M.D.,Ph.D., Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park CH, Hur J, Lee SM, Lee JW, Hwang SH, Seo JS, Lee KH, Kwon WC, Kim TH, Choi BW; LOGIS Investigators. Lipiodol lOcalization for Ground-glass opacity mInimal Surgery: Rationale and design of the LOGIS trial. Contemp Clin Trials. 2015 Jul;43:194-9. doi: 10.1016/j.cct.2015.06.009. Epub 2015 Jun 18. PMID 26093953